CLINICAL TRIAL: NCT05135546
Title: Inhaled Recombinant Non-immunogenic Staphylokinase vs Placebo in Patients With COVID-19 - FORRIF Trial
Acronym: FORRIF
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No patients
Sponsor: Supergene, LLC (Industry)
Collaborators: Russian Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: FORRIF
Record Dates: First submitted 2021-11-24; First posted 2021-11-26 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: At clinical centers, patients will be randomly distributed by the "envelope method" into two groups to receive Fortelyzin® or placebo.
  The drugs will be administered after the signed informed consent. Fortelyzin® will be administered by inhalation of a dose of 15 mg.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients and study investigators will be blinded to subject treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Recombinant nonimmunogenic staphylokinase lyophilisate for preparation of a solution for inhaled administration, 5 mg (745,000 IU) complete with a solvent. 15 mg (2,235,000 IU) - 3 vials, regardless of body weight.
  Interventions: Drug: Recombinant nonimmunogenic staphylokinase
- Placebo control (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant nonimmunogenic staphylokinase — 15 mg of drug reconstituted in 6 ml of 0.9% solution of NaCl for inhalation Other Name: Fortelyzin®
  Arms: Experimental
Drug: Placebo — 6 ml of 0.9% solution of NaCl for inhalation
  Other Names: Saline solution
  Arms: Placebo control

SUMMARY:
Objective: to evaluate the tolerability, safety and efficacy of inhaled usage of the Recombinant Non-immunogenic Staphylokinase (Fortelyzin®) vs placebo in patients with COVID-19.

DETAILED DESCRIPTION:
Fortelyzin® (the active substance Forteplase) is a recombinant non-immunogenic staphylokinase with high fibrinselective thrombolytic activity. In a multicentre, randomised clinical trial in patients with ST-segment elevation myocardial infarction (FRIDOM), non-immunogenic staphylokinase was administered as a single intravenous bolus of 15 mg in all patients, regardless of bodyweight, and showed similar high reperfusion patency and fewer minor bleeding events compared with tenecteplase, as well as the absence of neutralising IgGs. Results of the multicentre, randomised clinical trial in patients with an acute ischaemic stroke (FRIDA) suggested that the non-immunogenic staphylokinase administrated as a single intravenous bolus of 10 mg in all patients within the 4-5 h after the onset of symptoms is non-inferior to alteplase. Mortality, symptomatic intracranial haemorrhage, and serious adverse events did not differ between treatment groups (Gusev EI, Martynov MYu, Nikonov AA et al. Non-immunogenic recombinant staphylokinase versus alteplase for patients with acute ischaemic stroke 4-5 h after symptom onset in Russia (FRIDA): a randomised, open label, multicentre, parallel-group, non-inferiority trial. Lancet Neurol. 2021; 20(9): 721-728).

Complex coagulation and hematologic abnormalities, including significantly elevated D-dimer and fibrin/fibrinogen values are the distinct features identified in severe SARS-CoV-2. In the list of antithrombotic therapy drugs in conjunction with anticoagulant and antiplatelet therapy in patients with COVID-19, published by Liverpool Drug Interactions Group, fibrinolytic therapy is also included.

So the main objectives of this study are to assess the tolerability, safety and efficacy of inhaled usage of fibrinolytic agent the recombinant non-immunogenic staphylokinase (Fortelyzin®) in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and over
* Clinical status according to the WHO scale - 6, 7, 8 and 9 points.
* Verified respiratory infection COVID-19 by real-time PCR (quantitative)
* Patient consent to use reliable contraceptive methods throughout the study and for 3 weeks after:

  * women who have a negative pregnancy test and use the following contraceptives: intrauterine devices, oral contraceptives, contraceptive patch, prolonged injectable contraceptives, double barrier method of contraception. Women who are not fertile can also take part in the study (documented conditions: hysterectomy, tubal ligation, infertility, menopause for more than 1 year);
  * men using barrier contraception. The study may also involve men who are not fertile (documented conditions: vasectomy, infertility)
* Availability of signed and dated informed consent of the patient to participate in the study.

Exclusion Criteria:

* Clinical status according to the WHO scale - 1, 2, 3, 4 and 5 points.
* Increased risk of bleeding:

  * extensive bleeding at the present time;
  * intracranial (including subarachnoid) hemorrhage at the present time.
* Lactation, pregnancy
* Known hypersensitivity to Fortelyzin®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Number of patients discharged from the hospital with clinical status according to the WHO Ordinal Scale For Clinical Improvement - 3 points or less | 28 days post randomization
  The efficacy is evaluated in terms of the number of patients discharged from the hospital with clinical status according to the WHO Ordinal Scale For Clinical Improvement - 3 points or less

SECONDARY OUTCOMES:
Number of patients discharged from the hospital with clinical status according to the WHO Ordinal Scale For Clinical Improvement - 3 points or less | 14 days post randomization
  The efficacy is evaluated in terms of the number of patients discharged from the hospital with clinical status according to the WHO Ordinal Scale For Clinical Improvement - 3 points or less
Hospital length of stay | 28 days post randomization
  The efficacy is evaluated in terms of the hospital length of stay
Number of ICU-free days | 28 days post randomization
  The efficacy is evaluated in terms of the number of ICU-free days
Number of ventilation-free days | 28 days post randomization
  The efficacy is evaluated in terms of the number of ventilation-free days
Number of oxygen support-free days | 28 days post randomization
  The efficacy is evaluated in terms of the number of oxygen support-free days
SpO2 level | 7, 14 and 28 days post randomization
  The efficacy is evaluated in terms of the SpO2 level

CONTACTS AND LOCATIONS:
Overall Officials: Sergey S. Markin, MD, PhD, Principal Investigator — LLC "SuperGene"
Locations (2):
- Russia (2):
  - City Clinical Hospital No.52, Moscow
  - N.V. Sklifosovsky Research Institute of Emergency Medicine, Moscow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gusev EI, Martynov MY, Nikonov AA, Shamalov NA, Semenov MP, Gerasimets EA, Yarovaya EB, Semenov AM, Archakov AI, Markin SS; FRIDA Study Group. Non-immunogenic recombinant staphylokinase versus alteplase for patients with acute ischaemic stroke 4.5 h after symptom onset in Russia (FRIDA): a randomised, open label, multicentre, parallel-group, non-inferiority trial. Lancet Neurol. 2021 Sep;20(9):721-728. doi: 10.1016/S1474-4422(21)00210-6. PMID 34418399